CLINICAL TRIAL: NCT05986838
Title: Effect of Laser Puncture Versus Ultraviolet Radiation on Women With Polycystic Ovarian Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- laser puncture group (Active Comparator): gallium Arsenide infrared (GaAlAs) laser, using a wavelength at 904nm with a Maximum power output is 150 mW and a power density at 0.417 W/cm2 as well as an energy density of 4 J/cm2 will be employed for 2 minutes on specific acupuncture points
  Interventions: Device: aser puncture; Drug: Metformin
- Ultraviolet treatment group (Active Comparator): The therapist will place the UV arc lamp at a height of 60 to 80 cm above the lower abdomen region, perpendicular to the skin. Each woman's lamp will be switched on and given an individual timer by the minimum effective dose
  Interventions: Device: ultraviolet radiatio; Drug: Metformin
- Metformin only group (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Device: aser puncture — laser puncture (3 sessions per week)
  Arms: laser puncture group
Device: ultraviolet radiatio — ultraviolet radiation (3 sessions per week)
  Arms: Ultraviolet treatment group
Drug: Metformin — for 3 months

SUMMARY:
Obese women with polycystic ovarian syndrome aged between 25 and 35 years old will be divided into three groups. For three months, group (A) will receive laser puncture (3 sessions per week), along with a metformin supplementation, group (B) will receive ultraviolet radiation (3 sessions per week), along with a metformin supplementation, while group (C) will receive only metformin supplementation. The follicular size will be measured using ultrasound, while, female sex hormones, and serum 25-hydroxyvitamin D levels will bel evaluated using blood analysis

DETAILED DESCRIPTION:
Obese women with polycystic ovarian syndrome aged between 25 and 35 years old will be divided into three groups. For three months, group (A) will receive laser puncture (3 sessions per week), along with a metformin supplementation, group (B) will receive ultraviolet radiation (3 sessions per week), along with a metformin supplementation, while group (C) will receive only metformin supplementation. The follicular size will be measured using ultrasound, while, female sex hormones, and serum 25-hydroxyvitamin D levels will bel evaluated using blood analysis

ELIGIBILITY:
Inclusion Criteria:

* Obese nulli gravid PCOS women
* BMI 30-40 kg/m2

Exclusion Criteria:

* hyperprolactinemia
* BMI > 40 kg/m2 Endocrinological disorders such as thyroid disease, Cushing's syndrome, Coagulopathy
* Recent use of oral contraceptive pills
* Recent use of any photosensitizing medications, such as aspirin, tetracycline, chlorothiazide, or psoralen suspicious of neoplasms

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
LH/FSH ratio | 1 month after treatment
  LH/FSH ratio measured in venous sample on day 3 of the menstrual cycle

SECONDARY OUTCOMES:
Serum 25-hydroxyvitamin D concentration | 1 month after treatment
  25-hydroxyvitamin D measured in venous sample

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Maged, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No